CLINICAL TRIAL: NCT06127758
Title: The Effect of Virtual Reality Glasses Application on Surgical Fear and Anxiety in Patients Planned for Open Heart Surgery
Brief Title: Effect of Virtual Reality Glasses Application on Surgical Fear and Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, sabriye gül, postgraduate student, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0031
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Virtual Reality; Fear; Anxiety State; Surgery
Keywords: Heart surgery; surgical fear; anxiety; virtual reality
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VRG (Experimental)
  Interventions: Other: virtual reality glasses application; Other: classical training
- control group (Active Comparator)
  Interventions: Other: classical training

INTERVENTIONS:
Other: virtual reality glasses application — The experimental group will be given classical training (how to perform the surgery, complications that may occur after the surgery, preparation of fresh blood on the day of surgery, shaving by the barber on the morning of the surgery, how to take care of the mouth after shaving, how to shower with chlorexidine sponges, use of an apron, cap and mask after the shower). After 15 minutes video containing nature images and sounds will be shown through virtual glasses.
  Arms: VRG
Other: classical training — Information about classical training (how to perform the surgery, complications that may occur after the surgery, preparation of fresh blood on the day of surgery, shaving by the barber on the morning of the surgery, how to take care of the mouth after shaving, how to shower with chlorexidine sponges, use of an apron, cap and mask after the shower) will be given.

SUMMARY:
Purpose and Type of Research:This study will be conducted to examine the effect of virtual reality glasses on surgical fear and anxiety in patients scheduled for cardiovascular surgery. The study is a randomized controlled experimental research.

Method:The population of the research was approximately 2900 patients who underwent cardiovascular surgery in a year at Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Education Research Hospital. The sample size of the study was calculated using the G*Power software program.The study will be completed with 60 people by taking 30 people into the experimental and control groups.Data will be collected with a personal information form, surgical fear scale and state anxiety scale.

Hypothesis of the Research:

H1: Application of virtual reality glasses reduces surgical fear in patients planned for cardiovascular surgery.

H2: Application of virtual reality glasses reduces anxiety in patients scheduled for cardiovascular surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Those who will undergo open heart surgery,
* Those who have not had cardiovascular surgery before,
* No communication problems,
* Is conscious and able to answer questions and does not have any disorder/disease that affects decision-making ability (dementia, Alzheimer's, etc.),
* Does not have a psychiatric disease such as anxiety disorder, panic attack, depression,
* Individuals who do not receive psychiatric treatment such as antipsychotics/anxiolytics will be included in the study.

Exclusion Criteria:

* Being under the age of 18,
* Not having open heart surgery,
* Those who have previously undergone cardiovascular surgery,
* Having communication problems,
* Those who are unconscious and unable to answer questions Having any disorder/disease that affects decision-making ability (dementia, Alzheimer's, etc.),
* Having a psychiatric disease such as anxiety disorder, panic attack, depression,
* Individuals receiving psychiatric treatment such as antipsychotic/anxiolytic will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Personal Information Form | for 1 day
  The form prepared by the researchers contains a total of 8 questions containing the patients' introductory information.
surgical fear scale | for 1 day
  There are 8 questions in the scale. The scale is an 11-point Likert type scale with a score between 0 and 10. The scale included two subscales related to the source of fear, each consisting of 4 items. While items 1 to 4 on the scale measure the fear of the short-term consequences of surgery, items 5 to 8 measure the fear of the long-term consequences of surgery (0: not at all afraid, 10: very afraid). An increase in the score indicates an increase in fear.
state anxiety scale | for 1 day
  It consists of a total of 40 items and is scored from 1 to 4. Scale items are evaluated using the "Likert type" scaling method as "1 = not at all", "2 = a little", "3 = a lot", "4 = completely". A high score on the scale indicates a high level of anxiety; A low score indicates a low level of anxiety. In the validity and reliability study of the scale, the alpha value was found to be 0.91.

IPD SHARING:
Plan to Share IPD: No